CLINICAL TRIAL: NCT05475899
Title: Comparison of Instrument Assisted Soft Tissue Mobilization and Kinesiology Taping on Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/01048 Sidra Tariq
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Plantar Fascitis
Keywords: Plantar fasciitis; Instrument assisted soft tissue mobilization.; kinesiology taping
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instrument assisted soft tissue mobilization (Active Comparator): Patients in group A will be treated with the help of Instrument Assisted soft tissue mobilization GRASTON technique along with the conventional treatment. • Patient will be prone position with the foot over the edge of the table. Instrument will be applied from downward to upward direction with maximum of 10 - 15 strokes per session. These strokes will be applied in two sets of 10 strokes followed by stretches after each set. Conventional treatment includes icing and stretching of the calf muscles. Icing will be done for the total of 3-5 minutes. Both groups will be given session of 40 min/day, 3 days/week for 4 weeks, assessment will be done at baseline, at the end of 2nd week & at the end of 4th week.
  Interventions: Device: Instrument assisted soft tissue mobilization
- kinesiology taping (Experimental): Patients in group B will be treated with the help of kinesiology taping along with the conventional treatment. Patient will be in prone position with the dorsiflexion of the foot supported on the bed. Fan shaped taping will be applied with 60 - 100 % tension in the centre of the tape. The ends of the tape; the anchor will be applied without any stretch while centre of the tape will be stretched to approximately 60 - 100 %. Length of the tape may vary from person to person depending upon the size of the foot. Patient will be instructed to keep the tape till the next session. Conventional treatment includes icing and stretching of the calf muscles. Icing will be done for the total of 3-5 minutes. Both groups will be given session of 40 min/day, 3 days/week for 4 weeks, assessment will be done at baseline, at the end of 2nd week & at the end of 4th week.
  Interventions: Device: Instrument assisted soft tissue mobilization

INTERVENTIONS:
Device: Instrument assisted soft tissue mobilization — Application of IASTM on the plantar fascia with 10-15 strokes followed by stretching
  Other Names: Conventional Treatment: cold pack and Stretching exercises

SUMMARY:
The main objective of this study is to compare the effects of Instrument Assisted soft tissue mobilization and kinesiology taping on the pain, disability and range of motion of the patients and to compare the cost-effectiveness of both these treatment approaches. RCT done at health professionals, Life Care International hospital, and railway general hospital. The sample size was 36. Patients diagnosed with plantar fasciitis were randomized into 2 groups i.e., Group A and Group B with the help of non-probability convenience sampling. Both groups had received conventional Physiotherapy interventions (Stretching, Manual therapy, exercise therapy and home exercise plane.) along with specific techniques. The patients in group A had received Instrument assisted soft tissue mobilization (IASTM) and patients in group B had received treatment with kinesiology taping. The total duration of study was about 4 weeks. The patients had received 3 sessions per week for a period of 4 weeks and the outcomes were evaluated at baseline (first session), second assessment at the end of 2nd week and 3rd assessment at the end of 4th week. Only obese patients aged between 25-65 years were included in the study and were assessed upon the scoring of foot function index. Data will be analysed with the help of SPSS version 21.

DETAILED DESCRIPTION:
Plantar fasciitis is a common overuse injury that occurs as a result of repetitive traction forces on the plantar fascia at its origin over the distal calcaneus. Patients will complain of plantar heel pain, which is sharp rather than dull & exacerbated with the first step after a period of non-weight-bearing, typically in the morning. Plantar fasciitis is characterized by classic signs of inflammation including pain, swelling and loss of function but some presentations of plantar fasciitis may be a non-inflammatory. Pain is usually worse when barefoot on hard surfaces and with stair climbing. Pain relievers with walking initially & by stretching of longitudinal arch because Achilles' tendon is tight & dorsiflexion is limited.

The average plantar heel pain episode lasts longer than 6 months and it affects up to 10-15 % of the population. However, approximately 90 % of cases are treated successfully with conservative care. It is estimated that 1 in 10 people will develop PF during their lifetime. PF, which is more common in middle-aged obese females and young male athletes, has a higher incidence in the athletic population though not all suffering requires medical treatment. It is thought to occur in about 10 % of the general population as well, with 83 % of these patients being active working adults between the ages of 25 and 65 years old. Plantar fasciitis is diagnosed on the basis of medical history and physical examination including inspection and palpation to check for inflammation and tenderness.

Plantar fasciitis is defined as a localized inflammation & degeneration of planter fascia (a thick, broad, inelastic band of fibrous tissue on the plantar surface). The most widely accepted diagnostic test for plantar fasciitis is windlass test. It is performed by passively dorsiflexing the big toe of the involved foot in either weight bearing or non-weight bearing condition. Test will be positive when patient feels pain on the plantar surface while dorsiflexing the big toe. Treatments of plantar fasciitis include pharmacological therapy [medications (oral analgesics such as acetaminophen and nonsteroidal anti-inflammatory drugs) , injections (local anesthetics, steroids, botulinum toxin A, and/or saline)] Physiotherapy (Gastrocnemius-soleus stretching , dry needling, IASTM (instrument assisted soft tissue mobilization), extracorporeal shock wave therapy, exercise therapy, ultrasound therapy, iontophoresis, laser therapy, splints and kinesiology taping), and Surgery (fasciotomy, cryosurgery) Taping is beneficial technique for planter fasciitis in short term treatment & can be implemented as an immediate pain reliever. It helps in pain reduction, joint support, proprioception & muscle tone normalization. It has immediate positive effect on pain & function. The use of kinesiology taping results in better functional performance & balance. It has reduced pain in patients who use it as a short-term treatment. One intervention growing in popularity is Kinesio Tape and is marketed to be an easy-to-use, easily accessible, and cost-effective treatment option. Several theories have been proposed to describe its effect. The most widely-accepted theory states that the tape simulates the elasticity of skin and serves to pull the outer layer of skin off the underlying muscle and soft tissue structures, improving muscle function and decrease pressure on soft tissues, and create a larger space and channel for enhanced lymph flow . Another study in 2018 to check the effectiveness of kinesiology tape in plantar fasciitis. The study was an experimental study. Forty subjects were randomly allocated into two groups - Taping and control groups. The taping group (KT group) consisted of 20 subjects and intervened with the application of kinesiology tape (K tape). The control group consisted of 20 subjects and plantar fascia and calf stretching exercises were given during the treatment period. The results showed that the experimental group had a significant improvement in functional performance and dynamic balance when compared to the control group. Both male and female subjects in the age group of 40 to 60 years, subjects presenting with the symptoms of plantar fasciitis for more than 6 months were included. I have selected kinesiology taping for my study because I want to explore about it effects on subacute and chronic patients and to compare its cost effectiveness with other treatments available for this condition.

Instrument assisted soft tissue mobilization is a popular treatment for myofascial restriction. IASTM uses specially designed instruments to provide a mobilizing effect to scar tissue and myofascial adhesions. Several IASTM tools and techniques are available such as the GRASTON ® technique. A study was conducted to determine the effectiveness of GRASTON Technique® for decreasing pain and increasing function in participants with chronic plantar heel pain over a six-week period. A single blind, was conducted with a sample of 22 adults (5 males, 17 females). Participants were assigned to three groups: GT/stretching, effleurage/stretching, and stretching only. Participants improved in variables measured over a six-week treatment of GT. I have selected GRASTON technique in comparison with kinesiology taping in order to check which is most effective in terms of cost and treatment approach and to see in how many sessions patients with subacute and chronic plantar fasciitis will get results.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participants falling in this category will be recruited into the study.
* Patients with subacute and chronic plantar fasciitis.
* Positive windlass test (Aggravation of pain with passive dorsiflexion of big toe, during walking and standing on toes). Patients with a minimum FFI (pain and disability) rating score of 4. Pain worse on the first few steps in the morning.
* Both males and females
* Obese patients.
* Active working adults between the ages of 25 and 65 years old
* Patients who agreed not to wear high heeled shoes during study.

Exclusion Criteria:

* Patients having any other medical condition or trauma
* Patients sensitive to any of the above mentioned treatment modalities.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Foot function index (FFI) | 2nd week.
  It is a 23 scale measure instrument which is divided into 3 categories of pain, disability and activity limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Affan Iqbal, PhD*, Principal Investigator — Riphah International University
Locations (2):
- Pakistan (2):
  - Life care International hospital, Rawalpindi, Punjab Province
  - The Health Professionals, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No